CLINICAL TRIAL: NCT03099070
Title: Acute Stress Response in Migraine Sufferers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was severely delayed during COVID, and Grant support ended
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy Houle, Associate Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P001834
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Migraine Headache
Keywords: Stress; Fasting; Migraine
MeSH Terms: conditions — Migraine Disorders; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: 2 x 2 randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control, Not-Fasting (No Intervention): Participants will experience the control intervention and will not fast prior to the lab visit.
- Control, Fasting (Experimental): Participants will experience the control intervention and will fast prior to the lab visit.
  Interventions: Other: Fasting
- Stress, Not-Fasting (Experimental): Participants will experience the stress intervention and will not fast prior to the lab visit.
  Interventions: Behavioral: Stress
- Stress, Fasting (Experimental): Participants will experience the stress intervention and will fast prior to the lab visit.
  Interventions: Behavioral: Stress; Other: Fasting

INTERVENTIONS:
Behavioral: Stress — Trier Social Stress Test
  Arms: Stress, Fasting; Stress, Not-Fasting
Other: Fasting — 12-hour fasting prior to study visit
  Arms: Control, Fasting; Stress, Fasting

SUMMARY:
This study will examine the influence of stress and fasting on headache activity. Participants will receive both a control and stress session and be randomized to either fasting or not fasting for the visits.

DETAILED DESCRIPTION:
Stress and headache are intricately interrelated. Stress is thought to contribute to headache disorder onset in predisposed individuals, trigger or worsen individual headache episodes in those with headache, and exacerbate the progression of a headache disorder. In exacerbating headache disorder progression, stress is believed to be a major factor in headache transformation from an episodic to a chronic condition.

Broadly stated, stress is conceptualized as an imbalance between a demand, whether actual or perceived, and resources to handle the demand, resulting in a strain on the system. A stressor is any challenge or threat, whether objectively verified or not, to normal functioning. The stress response is the body's activation of physiological systems to protect and restore functioning.

This study is 2 x 2 experiment using male and female migraine sufferers. Participants will be randomized to a fasting or not fasting condition for the visits. Thus, the experiment is a 2 (control versus stress) x 2 (fasting versus not). During the approximately 4 weeks of participation (ranging from 9 to a maximum of 28 days), a participant also will complete a twice-daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18-65 years of age
* A provisional diagnosis of migraine (with or without aura).
* Headache frequency of 2 to 15 attacks/month

Exclusion Criteria:

* Presence of a secondary headache disorder (e.g., brain tumor)
* Chronic daily headache (> 15 headache days/month) or medication over-use headache (> 8 abortive medication doses/month)
* Recent change in nature of headache symptoms over last 6 weeks
* Not being able to read or speak English at a 6th grade level
* Any condition that would preclude the safe experience of a benign laboratory stressor including seizure disorder, Axis-I psychotic disorder, unstable cardiac conditions
* An active substance dependence issue (e.g., alcohol, marijuana) that interferes with data collection and headache activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Headache/Medication Use | Duration of lab visit (6 hours)
  The presence of a headache attack that is >= 4/10 on a 0 to 10 scale or a headache attack that requires the use of abortive/analgesic medication

SECONDARY OUTCOMES:
Time to next headache attack | 48 hours
  Time-to-event analysis using diary information
Medication use | 48 hours
  Frequency of abortive/analgesic medication use
Pain Scores | 6 hours
  Intensity of pain ratings (0 to 10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy T Houle, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No